CLINICAL TRIAL: NCT07286513
Title: A Prospective, Multi-Center Post-Market Clinical Study Evaluating the Safety, Performance, and Clinical Benefits of the Persona® SoluTion® PPS Femur
Brief Title: Persona SoluTion PPS Femur PMCF
Status: Not yet recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2025-04K
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Rhematoid Arthritis; Osteo Arthritis of the Knee; Traumatic Arthritis of Knee (Diagnosis); Polyarthritis; Collagen Disorders; Avascular Necrosis of Femoral Condyle; Valgus Deformity; Varus Deformity; Flexion Deformity of Knee
Keywords: Total Knee; Total knee arthroplasty; Knee replacement
MeSH Terms: conditions — Disease; Arthritis; Collagen Diseases | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will take a blood draw for a metal -Lymphocyte Transformation Test (metal-LTT) test to be performed by Orthopedic Analysis, LLC.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Persona® SoluTion PPS CR Femur with MC Bearing, cementless: This cohort will consist of subjects who receive the Persona® SoluTion PPS Cruciate Retaining Femur with the Medial Congruent Bearing, with cementless fixation.
  Interventions: Device: Total knee arthroplasty
- Persona® SoluTion PPS PS Femur with PS Bearing, cementless: This cohort will consist of subjects who receive the Persona® SoluTion PPS Posterior Stabilized Femur with the Posterior Stabilized Bearing, with cementless fixation.
  Interventions: Device: Total knee arthroplasty
- Persona® SoluTion PPS CR or PS Femur, cemented: This cohort will consist of subjects who receive the either the Persona® SoluTion PPS Cruciate Retaining Femur (with the Medial Congruent Bearing) or Posterior Stabilized Femur (with the Posterior Stabilized Bearing), with cemented fixation.
  Interventions: Device: Total knee arthroplasty

INTERVENTIONS:
Device: Total knee arthroplasty — The screening population will consist of patients for whom clinical decision has been made to use the Persona® SoluTion® PPS femoral implant in total knee arthroplasty prior to enrollment in the research.
  Other Names: Total Knee replacement

SUMMARY:
The goal of this study is to generate clinical evidence and evaluate the safety and performance of the Persona® SoluTion® PPS Femurs in the US market, with data supporting global regulatory submissions, including CE marking under EU MDR.

The target population consists of adults undergoing knee arthroplasty with the Persona SoluTion femoral component paired with a Medial Congruent (MC) or Posterior Stabilized (PS) articulating surface in line with its current cleared Instructions for Use (IFU).

The primary endpoint is the assessment of clinical performance and benefits by evaluating the average change in the KOOS JR score between pre-operative and 2-year post-operative follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is of legal age of consent and skeletally mature
2. Patient is willing and able to provide written Informed Consent by signing and dating the IRB/EC approved Informed Consent document
3. Patient is willing and able to complete scheduled follow-up evaluations as defined in the study protocol
4. Patient qualifies for total knee arthroplasty based upon physical exam and medical history and meets the approved indications for use of the Persona® SoluTion® PPS femoral implant and appropriate compatible components, within a pre-specified variant configuration (cohort).
5. A clinical decision has been made to use the Persona® SoluTion® PPS femoral implant prior to enrollment in the research

Exclusion Criteria:

1. Patient is currently participating in any other surgical intervention or pain management study
2. Patient is pregnant or considered a member of a protected (vulnerable) population whose inclusion in the study is inappropriate (e.g. prisoner, mentally incompetent)
3. Patient has a mental or neurologic condition who is unwilling or incapable of following postoperative care instructions
4. Patient has a condition which would, in the judgement of the Investigator, place the patient at undue risk or interfere with the conduct of the study
5. Patient is institutionalized or is a known drug abuser, a known alcoholic or cannot understand the requirements of study participation
6. Previous history of infection in the affected joint and/or other local/systematic infection that may affect the prosthetic joint
7. Insufficient bone stock on femoral or tibial surfaces
8. Skeletal immaturity
9. Neuropathic arthropathy
10. Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
11. A stable, painless arthrodesis in a satisfactory functional position
12. Severe instability secondary to the absence of collateral ligament integrity
13. Rheumatoid arthritis (RA) accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
14. Study device not implanted during surgery, or surgery did not occur
15. KOOS JR score not collected pre-operatively
16. Patient requires simultaneous bilateral knee surgery for treatment of the diagnosed condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should be a consecutive series of subjects implanted with the Persona® SoluTion® PPS Femurs along with the corresponding Vivacit-E polyethylene articulating surface that meet the inclusion and exclusion criteria. To avoid selection bias, each Investigator will prospectively offer study participation to each consecutive potential and eligible patient for primary TKA using the commercially available Persona® SoluTion device. Bilateral patients requiring simultaneous surgical treatment will not be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Change in KOOS JR Score between pre-op and 2 years post-op | 2 years
  A 7-item shortened version of the Knee injury and Osteoarthritis Outcome Score (KOOS), specifically designed to assess knee health in patients undergoing total knee arthroplasty (TKA). Raw scores are converted to an interval score ranging from 0 to 100, where 0 represents complete knee disability and 100 represents perfect knee health (higher scores indicate less pain and better function).

SECONDARY OUTCOMES:
KOOS JR Score | 5 years
  A 7-item shortened version of the Knee injury and Osteoarthritis Outcome Score (KOOS), specifically designed to assess knee health in patients undergoing total knee arthroplasty (TKA). Raw scores are converted to an interval score ranging from 0 to 100, where 0 represents complete knee disability and 100 represents perfect knee health (higher scores indicate less pain and better function).
Oxford Knee Score (OKS) | 5 years
  A 12-item PROM was specifically designed and developed to assess function and pain after TKA. This tool is short, reproducible, valid, and sensitive to clinically important changes. Possible scores range from a minimum 0 to maximum 48 points, with higher scores indicating less pain and fewer functional limitations.
EuroQol-5 Dimension-5 Level (EQ-5D-5L) Questionnaire | 5 years
  The EQ-5D-5L instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS). The questionnaire produces an "index" score that ranges from 0 to 1, where 0 is the value of a health state equivalent to dead; and 1 is the value of full health, with higher scores indicating higher health utility. The EQ VAS is a 0 -100 scale where patients are asked to indicate their overall health on the day of questionnaire completion. 100 indicates the best health imaginable and 0 indicates the worst health imaginable. Change in Index and EQ VAS scores will be compared from baseline to 2-year follow-up as well as from baseline to 5-year postoperative follow-up for each cohort. This change will also be compared between the cohorts.
Numeric Rating Scale (Pain) | 5 years
  The 11-item pain NRS asks patients to rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"). It is the most widely used instrument for pain screening with higher scores indicating greater pain intensity.
Survival Rate of Implant | 10 years
  Survival Rate (Survivorship) will be both assessed by revision/additional surgeries to the affected joint due to aseptic loosening only or by revision, removal, exchange of the implanted device due to any reason. Aseptic loosening and other reasons for additional surgeries may be identified by radiographic imaging.
Frequency and types of Adverse Events | 10 years
  The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.
Assessment of the prevalence of metal hypersensitivities using a metal Lymphocyte Transformation Test (LTT) | 10 years
  The Orthopedic Panel 2 tests for hypersensitivity to aluminum, cobalt, chromium, iron, molybdenum, nickel, vanadium, zirconium, titanium alloy particles, cobalt alloy particles, bone cement particles, and bone cement liquid.

OTHER OUTCOMES:
Patient Expectations Pre- and Post-op | 5 years
  Per the 2011 Knee Society scoring manual: "[This] is a three-question fifteen-point scale that is collected pre-operatively and post-operatively. The pre-operative questions reflect the patient's opinion on the extent to which the patient expects that the operation will improve their knee pain, and their ability to perform their activities of daily living and recreational activities. The post-operative questions reflect the extent to which the outcome after the operation has met the patient's pre-operative expectations with respect to pain and function." Higher scores preoperatively indicate more positive expectations of the patient's total knee replacement surgery, and higher scores postoperatively indicate the level to which a patient's pre-op expectations have been met.
Patient Satisfaction Questionnaire | 5 years
  A three-question Patient Satisfaction Questionnaire. The questions include general satisfaction, level of pain, and a hypothetical question about whether the patient would do the surgery again.
Assessment of Radiographic Outcomes | 10 years
  Radiographic parameters to be evaluated include, but are not limited to, radiolucencies, osteolysis, hypertrophy, subsidence, and heterotopic ossification. All radiographic evaluations performed according to the protocol will be reviewed by the investigator at the time of the evaluation for significant radiographic findings.

IPD SHARING:
Plan to Share IPD: Undecided